CLINICAL TRIAL: NCT07106879
Title: Pre-screening Survey for Metabolic, Cardiovascular, Obesity, Mental Health, and Endocrine Trial Eligibility (DOVE-MET-COME-100)
Brief Title: Non-interventional Pre-screening Protocol Aims to Evaluate Participants for Potential Trial Eligibility in Future Clinical Trials/Studies Focusing on Metabolic and Psychiatric Health.
Status: Recruiting | Type: Observational
Sponsor: Clindove Research LLC (Other)
Responsible Party: Sponsor
Other Study IDs: METCOME062025
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome; Obesity; Prediabetes; Mental Health Disorders; Endocrine Dysfunction; Type 2 Diabetes Mellitus (T2DM); Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Obesity; Prediabetic State; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants undergoing metabolic and/or psychiatric assessments through blood work and structured clinical evaluations, as outlined in the study protocol.
  Interventions: Other: Blood Work

INTERVENTIONS:
Other: Blood Work — Collection of blood samples for metabolic and other necessary biomarker analysis, including Hemoglobin A1c (HbA1c), Lipid Panel, Liver and Kidney function tests and other protocol-defined assays.

SUMMARY:
DOVE-MET-COME-100 is a single site prescreening survey study designed to identify adults who may be eligible for future industry-sponsored clinical trials. A physician will oversee the informed consent process, after which participants will be surveyed on demographics, medical history, current health conditions and symptoms. The study team may also collect basic health information, including vital signs, urine drug tests, blood samples and pregnancy tests (if applicable). A physician will review each participant's medical history in a one-on-one interview to assess potential fit for upcoming trials. If needed, the doctor may contact the participant's current doctors or pharmacies to gather more information for eligibility review.

DETAILED DESCRIPTION:
Eligible participants will undergo screening procedures including laboratory assessments and health questionnaires to determine their suitability for further evaluation in metabolic and/or psychiatric sub-studies. The study does not include any investigational intervention.

ELIGIBILITY:
Inclusion Criteria:

* Any participant of age 18 years and over
* Who are willing to provide informed consent and participate in the pre-screening study and comply with study procedures.

Exclusion Criteria:

* Pregnant or breastfeeding individuals
* Individuals having severe cognitive impairment or inability to provide informed consent
* Individuals having acute psychiatric emergencies requiring immediate intervention/hospitalization
* Individuals who are currently participating in another research study that conflicts with pre-screening data collection
* Individuals having known history of drug/alcohol misuse
* Individuals having medical conditions that, in the investigator's opinion, could compromise the integrity of the screening process or pose significant risks to the participant's health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll participants of any sex, aged 18 and over from a general outpatient population, including both self-referred individuals and those referred by healthcare providers. Participants will undergo metabolic and/or psychiatric evaluations through structured interviews and blood-based biomarker assessments. Individuals interested in participating in an industry-sponsored clinical trial for investigational products targeting cardiovascular, obesity, or endocrine conditions will be screened for clinical suitability. Eligible participants may present with symptoms related to metabolic or psychiatric conditions, or both.
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who express interest in industry-sponsored clinical research | 5 years
  The number of participants who express interest in industry-sponsored clinical research in each of the following therapeutic areas: cardiovascular, endocrine, metabolic and mental health disorder.

SECONDARY OUTCOMES:
Development of a systematically curated and structured electronic database of pre-screened individuals, annotated with metabolic, cardiovascular, endocrine, and psychiatric risk factors | 5 years
  Development of a systematically curated and structured electronic database of pre-screened individuals, annotated with metabolic, cardiovascular, endocrine, and psychiatric risk factors, for the purpose of streamlined matching and recruitment into future interventional trials. This will include demographic, clinical, laboratory, and mental health data with longitudinal tracking capacity for re-contact and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Cohen, MD, Principal Investigator — Clindove Research LLC
Locations (1):
- Clindove Research LLC, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clindove Research LLC Website — https://clindove.com/

DOCUMENTS (1):
  • Informed Consent Form (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT07106879/ICF_000.pdf